CLINICAL TRIAL: NCT00837616
Title: Estrogen Dosing in Turner Syndrome:Pharmacology & Metabolism
Brief Title: Estrogen Dosing in Turner Syndrome: Pharmacology and Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nelly Mauras, Chief, Division of Endocrinology, Diabetes & Metabolism, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 908-M01
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Turner Syndrome; Hypogonadism; Premature Ovarian Failure
Keywords: Turner Syndrome; Hypogonadism; GH; Estrogen; Estrogen Patches; IGF-I; Body Composition; Protein Metabolism; Lipid Oxidation; Estradiol assay by LCMSMS; Recombinant Cell Bioassay
MeSH Terms: conditions — Turner Syndrome; Hypogonadism; Primary Ovarian Insufficiency | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A will receive the oral estradiol for 12 months
  Interventions: Drug: 17 B estradiol orally
- Group B (Active Comparator): Group B will receive the transdermal estradiol for 12 months
  Interventions: Drug: 17 B estradiol

INTERVENTIONS:
Drug: 17 B estradiol orally — Group A will be given estrogen by mouth daily(0.5 mg or 1mg or 2 mg of 17B Estradiol. Doses will vary depending on the blood levels of estrogen starting with the lower doses and adjusting these doses up as needed to keep the levels in the normal range. The estrogen will be taken for 21 days. In order to have a menstrual cycle progesterone will be given for 7 days, starting from day 14 through day 21 of each cycle. Then both medications are stopped on day 21 for a total of 7 days. Labs will be obtained at baseline, 1,2,3,6,9 and 12 months. Dual-energy X-ray absorptiometry (DXA) scan and calorimetry will be done at baseline and at 6 and 12 month.
  Other Names: Estrace
  Arms: Group A
Drug: 17 B estradiol — Group B will be given estrogen via a patch applied to the skin twice a week (0.375mg or 0.05mg or 0.075mg) Doses will vary depending on the blood levels of estrogen starting with the lower doses and adjusting these doses up as needed to keep the levels in the normal range. The estrogen will be taken for 21 days. In order to have a menstrual cycle progesterone will be given for 7 days, starting from day 14 through day 21 of each cycle. Then both medications are stopped on day 21 for a total of 7 days. Labs will be obtained at baseline, 1,2,3,6,9 and 12 months. Dual-energy X-ray absorptiometry (DXA) scan and calorimetry will be done at baseline and at 6 and 12 month.
  Other Names: Vivelle
  Arms: Group B

SUMMARY:
Estrogen is necessary for feminization during puberty and to decrease bone resorption, the latter critical for the achievement of peak bone mass and normal bone health in the female. The practicing pediatric endocrinologist often faces the dilemma of how to best feminize girls with hypogonadism (lack of estrogen), manifested as delayed or arrested puberty, due to disorders of the brain or the ovaries. We propose a series of studies to address which type, dose, and route of delivery of estrogen are suitable choices in feminizing and sustaining estrogen concentrations in adolescent girls with Turner syndrome. To accomplish this we will study girls/young woman between the ages of 13 to 20 with Turner Syndrome in 2 protocols. In Protocol # 1 we will study 24 girls with TS, they will receive 3 different estrogen preparations, either by mouth or via a patch for a total of 6 weeks. They will come to the clinical research center for blood draws after 2 wks of taking the estrogen. With this study, we hope to learn how the body responds to estrogen differently, depending on the form estrogen is given and how high, estrogen levels gets in the blood in these girls with Turner Syndrome. We will be comparing these patients estrogen levels to girls that menstruate normally and do not have Turner Syndrome. In Protocol #2, 40 patients with TS will be recruited; these patients will take estrogen for 1 year, either by mouth or via a patch. Patients will come to the lab for blood drawn in 7 occasions and we will measure estrogen levels as well as other hormones and lipid levels. We will also perform a Dual-energy X-ray absorptiometry (DXA) study (like an X ray) to assess body composition and bone mineralization. We will adjust doses based on the estrogen levels we find. With this study we hope to learn how estrogen affects body composition, i.e., the amount of fat vs. muscle, and how different forms of estrogen affect blood cholesterol and other hormones. This study will allow us to understand better how to best replace young woman with Turner Syndrome with estrogen.

DETAILED DESCRIPTION:
Data on the specific effects and bioequivalency of the different forms of estrogen are lacking, and in the young adolescent age group in particular, virtually non-existent. This has been complicated further by the difficulty in accurately interpreting estradiol assay results as the conventional radioimmunoassays (RIA) for estradiol are inaccurate and insensitive measuring very small concentrations in plasma. There is wide variation in the types of estrogens used for estrogen replacement, as well as doses and route of administration. Girls with Turner syndrome (TS) represent an important case study for these issues as they have early primary gonadal insufficiency or failure many years before the achievement of peak bone mass. Hence, a study of the effects of different estrogen compounds in this patient population offers a unique model that eliminates the confounding effects of other products produced by the intact gonad. Since in this condition it is imperative that estrogen replacement is started during the adolescent years and continued for several decades, this issue becomes highly relevant to these young women's health.Our specific aims are to: 1. to characterize the pharmacokinetics (PK) and pharmacodynamics (PD) and relative biological potency of different oral vs. transdermal preparations of estradiol using state-of-the-art tandem mass spectrometry assays and recombinant cell bioassays; 2. to investigate the differential, long term metabolic effects of oral vs. transdermal estrogen replacement, specifically the effects on lipid and protein metabolism as well as body composition in this patient population; 3. to determine feasibility of estrogen concentration-based dosing in puberty and 4. To characterize the metabolic profile of TS girls previously treated with GH. To accomplish this we will study girls/young woman between ages 13 to 20 with TS in 2 protocols. Protocol #1 will be a study of the pharmacokinetic/pharmacodynamic (PK/PD) of 3 different preparations of estrogen in different doses. Protocol #2 will be a one year longitudinal study of the effects of oral vs. transdermal (TD) estrogen on body composition, hormones and growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Girls with Turner Syndrome (45X, or related karyotypes) diagnosed clinically and cytogenetically
* Female subjects with Y material will be allowed providing gonadectomies have been performed previously
* Age: 13-20 years
* Subjects have completed or nearly completed their linear growth
* Previous growth hormone (GH) therapy discontinued at least 6 months prior to study participation
* Stable thyroid replacement therapy will be allowed
* Celiac disease on stable diets will be allowed
* Any previous hormone replacement therapy (HRT) will be allowed

Exclusion Criteria:

* Diabetes Mellitus on insulin therapy, insulin sensitizers or oral hypoglycemics
* Inflammatory Bowel Disease (ulcerative colitis or Crohn's disease), celiac disease
* Cigarette smoking
* Any other chronic conditions, that, in the opinion of investigators could impair the metabolism of nutrients
* Severe obesity, i.e., Body Mass Index (BMI) >95th centile

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (3):
- United States (2):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jefferson Medical College of Thomas Jefferson University, Philadelphia, Pennsylvania
- University of Chile/Clinica las Condes, Santiago, Chile

REFERENCES:
- [Result] Torres-Santiago L, Mericq V, Taboada M, Unanue N, Klein KO, Singh R, Hossain J, Santen RJ, Ross JL, Mauras N. Metabolic effects of oral versus transdermal 17beta-estradiol (E(2)): a randomized clinical trial in girls with Turner syndrome. J Clin Endocrinol Metab. 2013 Jul;98(7):2716-24. doi: 10.1210/jc.2012-4243. Epub 2013 May 15. PMID 23678038
- [Result] Taboada M, Santen R, Lima J, Hossain J, Singh R, Klein KO, Mauras N. Pharmacokinetics and pharmacodynamics of oral and transdermal 17beta estradiol in girls with Turner syndrome. J Clin Endocrinol Metab. 2011 Nov;96(11):3502-10. doi: 10.1210/jc.2011-1449. Epub 2011 Aug 31. PMID 21880799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-one girls with Turner Syndrome (45X and related karyotypes), between 13 and 20 years were recruited and followed among the 3 participating centers at the Nemours Children's Clinic, Jacksonville (coordinating center), Nemours Jefferson, and Clínica las Condes/University of Chile, Santiago, Chile.
Pre-assignment Details: Any previous growth hormone (GH) therapy was discontinued at least 6 months prior to study participation. Estrogen replacement therapy was discontinued for at least 6 weeks prior to baseline studies. Subjects with significant obesity (BMI > 36 kg/m2) or history of systemic illness were excluded.
Groups:
- Oral Estradiol: Group A received the oral estradiol for 12 months
- Transdermal Estradiol: Group B received the transdermal estradiol for 12 months
Period: Overall Study
Arm/Group | Oral Estradiol | Transdermal Estradiol
Started | 20 | 21
Completed | 20 | 20
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group A: Group A received the oral estradiol for 12 months
- Group B: Group B received the transdermal estradiol for 12 months
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (1.7) | 16.7 (1.8) | 16.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 25
  Chile | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
kilograms | 1.1 (0.6) | 1.9 (0.6)

2. Primary Outcome: Change in Body Mass Index From Baseline at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
kg/m2 | 0.075 (0.38) | 0.65 (0.38)

3. Primary Outcome: Change in Percent Fat Mass From Baseline in 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: percent fat mass
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
percent fat mass | -0.14 (0.56) | -0.64 (0.56)

4. Primary Outcome: Change in Fat Free Mass From Baseline at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
kg | 1.03 (0.37) | 1.67 (0.4)

5. Secondary Outcome: Changes in Insulin Growth Factor-I From Baseline at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
ng/ml | -16 (12) | 28 (12)

6. Secondary Outcome: Lipids Concentrations After Using Oral Versus Transdermal 17B Estradiol Replacement for 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
mg/dl
  Total Cholesterol | 168 (7) | 153 (6)
  Low Density Lipoprotein | 93 (4) | 88 (5)
  High Density Lipoprotein | 56 (3) | 50 (2)
  Triglycerides | 95 (19) | 70 (9)

7. Secondary Outcome: Rates of Lipid Oxidation After Using Oral Versus Transdermal 17B Estradiol Replacement for 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Kcal/Fat Free Mass/day
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
Kcal/Fat Free Mass/day | 10 (2.8) | 7.3 (1.6)

8. Secondary Outcome: Serum 17B Estradiol Concentrations After Using Oral Versus Transdermal 17B Estradiol Replacement for 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
pg/ml | 124 (19) | 74 (17)

9. Secondary Outcome: Serum Estrone Concentrations After Using Oral Versus Transdermal 17B Estradiol Replacement for 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
pg/mL | 504 (80) | 43 (7)

10. Secondary Outcome: Serum Estrone Sulfate Concentrations After Using Oral Versus Transdermal 17B Estradiol Replacement for 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Oral Estradiol | Transdermal Estradiol
Number analyzed (Participants) | 20 | 20
pg/mL | 63638 (21088) | 1875 (414)

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No